CLINICAL TRIAL: NCT02683044
Title: Randomized Clinical Trial To Evaluate The Comparative Effectiveness And Safety Of Two Protocols For The Treatment Of Erectile Dysfunction With Low-Density Shock Waves
Brief Title: Effectiveness And Safety Of Two Protocols For The Treatment Of Erectile Dysfunction With Low-Density Shock Waves
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto para la Evaluación de la Calidad y Atención en Salud (Other)
Collaborators: Boston Medical Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IECAS-BMG-01
Record Dates: First submitted 2016-02-09; First posted 2016-02-17 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-07

CONDITIONS: Erectile Dysfunction
Keywords: Erectile dysfunction; Low-Density Shock Waves; Randomized Clinical Trial
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Li-ESWT 5 weeks (Experimental): Consists of five sessions of Low-Intensity Extracorporeal Shock Wave Therapy , one per week, with 3000 pulses at 0,15 mg/mm2, at a frequency of 4 Hz. The distribution of the shocks will be 2000 pulses to the body of the penis and 1000 pulses at its base. Total duration: 5 weeks.
  Interventions: Procedure: Low-Intensity Extracorporeal Shock Wave Therapy (Li-ESWT)
- Li-ESWT 3 weeks (Active Comparator): Consists of six sessions of Low-Intensity Extracorporeal Shock Wave Therapy , two per week, with 1500 pulses each one at 0.1 mJ/mm2, at a frequency of 4 Hz. The distribution of the shocks will be 900 pulses to the body of the penis and 600 pulses at its base. Total duration: 3 weeks.
  Interventions: Procedure: Low-Intensity Extracorporeal Shock Wave Therapy (Li-ESWT)

INTERVENTIONS:
Procedure: Low-Intensity Extracorporeal Shock Wave Therapy (Li-ESWT) — Sessions of shocks to the body of the penis

SUMMARY:
Randomized, experimental, non-inferiority clinical trial to determine the comparative effectiveness and safety of two protocols used in the treatment of Erectile Dysfunction (ED) with Low-Density Shock Waves (Li-ESWT), for patients seen at the Boston Medical Group's Bogota center. Protocol 1: Consists of five sessions, one per week, with 3000 pulses at 0,15 mg/mm2, at a frequency of 4 Hz. The distribution of the shocks will be 2000 pulses to the body of the penis and 1000 pulses at its base. Total duration: 5 weeks. Protocol 2: Consists of six sessions, two per week, with 1500 pulses each one at 0.1 mJ/mm2, at a frequency of 4 Hz. The distribution of the shocks will be 900 pulses to the body of the penis and 600 pulses at its base. Total duration: 3 weeks.

Outcome variables: Erection Hardness Score (EHS). International Index of Erectile Function, 5-item version (IIEF-5). Penile blood flow.

Evaluation at 1, 3 and 6 months after completing each of the Li-ESWT protocols.

DETAILED DESCRIPTION:
Objectives

General

Determine the comparative effectiveness and safety of two treatment protocols for the use of low-intensity shock waves to treat patients with erectile dysfunction who are seen at the Boston Medical Group's Bogota center.

Specific

1. Determine differences in IIEF-5 and the EHS scores resulting from Li-ESWT therapy for patients with ED, upon completion of therapy and 1, 3 and 6 months thereafter, according to the type of protocol used.
2. Determine differences in penile blood flow resulting from Li-ESWT therapy for patients with ED, measured with doppler upon completion of therapy and 3 months thereafter, according to the type of protocol used.
3. Determine differences in adverse effects during Li-ESWT therapy for patients with ED, according to the type of protocol used.

Type of Study

Randomized, experimental, non-inferiority clinical trial to determine the comparative effectiveness and safety of two protocols used in the treatment of ED with Li-ESWT, for patients seen at the Boston Medical Group's Bogota center.

Investigation Hypothesis

Ho: Differences exist in the effectiveness of two treatment protocols for the use of Li-ESWT to treat erectile dysfunction, measured by an improvement in the EHS score one month after completing treatment.

Ha: No differences exist in the effectiveness of two treatment protocols for the use of Li-ESWT to treat erectile dysfunction, measured by an improvement in the EHS score one month after completing treatment.

Population

Patients diagnosed with ED who are treated at the Boston Medical Group's Bogota center. These patients must meet the eligibility criteria.

Sample Size

The sample size was calculated for non-inferiority, based on the new approach being at least as good as the existing one. The effectiveness of Protocol 1 is presumed to be 57%, according to the literature (12), and Protocol 2 is presumed to be least as good as Protocol 1. The difference in effectiveness between the two protocols should be less than or equal to 20%. With a power of 80% and a significance level of 97.5%, a one-tailed test requires a sample size of 97 individuals per arm. Since a maximum of 5% of patients are expected to be lost in the first month post-treatment, a final sample size of 103 individuals per arm was calculated and, therefore, a total of 206 individuals will be randomly assigned. These calculations are performed using the Stata 14© ssi module.

Interventions

Each patient will be randomly assigned to one of the two arms. The patients in each arm will be treated by one of the two protocols described below. These protocols will be administered by two Li-ESWT machines from either Storz Duollith, Medispec or MTS.

The protocols are:

* Protocol 1: Consists of five sessions, one per week, with 3000 pulses at 0,15 mg/mm2, at a frequency of 4 Hz. The distribution of the shocks will be 2000 pulses to the body of the penis and 1000 pulses at its base. Total duration: 5 weeks.
* Protocol 2: Consists of six sessions, two per week, with 1500 pulses each one at 0.1 mJ/mm2, at a frequency of 4 Hz. The distribution of the shocks will be 900 pulses to the body of the penis and 600 pulses at its base. Total duration: 3 weeks.

Outcome Variables

Effectiveness

The principal outcome variables with which the effectiveness of each intervention will be measured will be:

* Erection Hardness Score (EHS). The EHS has a single Likert scale, and the validated Spanish version will be used (27). The score is as follows: 0 = Penis does not increase in size; 1= the penis increases in size but is not hard; 2 = the penis is hard but not hard enough for penetration; 3 = the penis is hard enough for penetration but not completely hard; 4 = the penis is completely hard and fully rigid (Appendix 1).
* International Index of Erectile Function, 5-item version (IIEF-5). Five questions related to erectile function, orgasmic function, sexual desire, satisfaction with sexual relations and overall satisfaction. In addition, this has a high sensitivity and specificity for detecting changes in erectile function in response to treatment. The ED grade is scored on a scale of 0 to 25 points, where: 5-7 is severe, 8-11 is moderate, 12-16 is mild to moderate; 17-21 is average; and 22-25 ED does not exist (28) (Appendix 2).
* Penile blood flow with vasoactive stimuli of prostaglandin (VSP), measured by color echo-doppler. After applying a standard dosage of VSP, an exam measures blood flow in the cavernous and dorsal arteries at the base of the penis. This measurement is performed periodically every 5 minutes, as of the application of the medication until obtaining the best possible flow. This determines normal flow when above 35 cm/sec , undetermined when between 25 and 35 cm/sec and abnormal flow when under 25 cm/sec.

The scores from the EHS and IIEF-5 scales will be measured at baseline, upon completion of each protocol, and 1, 3 and 6 months after completing each protocol. Doppler measurements of penile arteries will be taken at baseline and 1 month after completing each protocol.

Safety

This will be determined according to the presence of adverse events, which will be analyzed upon completion of each therapy and after 1, 3 and 6 months (control months). This variable will be dichotomous, as the presence or absence of adverse events. It is important to emphasize that no adverse events have been reported to-date by any clinical trial of patients with ED who have been treated with Li-ESWT (12, 14, 19, 29).

Techniques, Procedures and Data Collection and Processing

Subjects who are seen for a private consultation at the Boston Medical Group's Bogota center will be screened to define whether they meet the eligibility criteria. If they are eligible they will be invited to participate in the investigation and will be given an informed consent form which explains the objectives of the investigation as well as the risks involved in participating in the study.

The patients will then be assigned to one of two arms through the process of selecting a ballot among a group of ballots marked with the protocols and stored in a dark bag. Prior to beginning the two protocols, a baseline measurement will be taken of the outcomes related to the study's objectives (EHS, IIEF-5 and doppler measurement of blood flow in the cavernous artery). In accordance with the results from the randomization process, each subject will be treated by one of the protocols mentioned in the corresponding section.

Upon completion of the administration of the protocols, EHS and IIEF-5 scores will be measured a second time, as well as any associated adverse effects. This will be done five weeks after beginning treatment for subjects in Protocol 1 and three weeks after beginning treatment for subjects in Protocol 2.

Medical check-ups will be performed by doctors who are experienced in the treatment of male sexual dysfunction. These will be conducted 1, 3 and 6 months after completing each of the Li-ESWT protocols. EHS and IIEF-5 scores will be determined at these consultations, as well as the presence or absence of adverse events related to the therapy. A second measurement of penile blood flow will be taken with doppler echography one month after completing each of the protocols.

All the information will be recorded in the electronic clinical history which already exists at the Boston Medical Group. The clinical information will be extracted from this electronic clinical history once all the data from the sample has been collected. This information will be exported to a flat file so it can be read later by a statistical package.

In terms of historical information, 4 to 5 individuals are expected to be included in the study per week. Based on this supposition, approximately 52 weeks will be needed for the inclusion of individuals. The last individual included will be followed up to the sixth month after completion of therapy.

Follow-up and Loss-to-Follow-up

One person involved in the project and a medical supervisor will be responsible for conducting a telephone follow-up of the patients included in the study. This will be done with the expectation of guaranteeing a loss-to-follow-up of under 5% in the first month post-therapy.

ELIGIBILITY:
Inclusion Criteria:

* Presence of ED for more than 3 months in over 50% of sexual intercourses.
* EHS score under or equal to 3.
* IIEF-5 score under or equal to 21.
* Patients who agree to participate in the trial through signed informed consent.

Exclusion Criteria:

* Active bladder, prostate or colon cancer.
* Patients with ED having a psychological origin.
* Any psychiatric pathology, spinal cord injury or anatomical penile dysfunction.
* Patients with INR over 3, ordered by a cardiologist.
* Patients with clinically suspected hypogonadism (AMS under 36).
* Patients with active infections or lesions on the penis or pubic area.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-08 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Erection Hardness Score (EHS) | 1 month after completing each protocol

SECONDARY OUTCOMES:
Penile blood flow | 1 month after completing each protocol
  Penile blood flow with vasoactive stimuli of prostaglandin (VSP), measured by color echo-doppler
International Index of Erectile Function, 5-item version (IIEF-5) | 1, 3 and 6 months after completing each protocol
Erection Hardness Score (EHS) | 3 and 6 months after completing each protocol

CONTACTS AND LOCATIONS:
Overall Officials: Jose P Saffon, MD, Principal Investigator — Boston Medical Group
Locations (1):
- Boston Medical Group, Bogotá, Bogota D.C., Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosen RC, Fisher WA, Eardley I, Niederberger C, Nadel A, Sand M; Men's Attitudes to Life Events and Sexuality (MALES) Study. The multinational Men's Attitudes to Life Events and Sexuality (MALES) study: I. Prevalence of erectile dysfunction and related health concerns in the general population. Curr Med Res Opin. 2004 May;20(5):607-17. doi: 10.1185/030079904125003467. PMID 15171225
- [Background] Lewis RW, Fugl-Meyer KS, Corona G, Hayes RD, Laumann EO, Moreira ED Jr, Rellini AH, Segraves T. Definitions/epidemiology/risk factors for sexual dysfunction. J Sex Med. 2010 Apr;7(4 Pt 2):1598-607. doi: 10.1111/j.1743-6109.2010.01778.x. PMID 20388160
- [Background] Braun M, Wassmer G, Klotz T, Reifenrath B, Mathers M, Engelmann U. Epidemiology of erectile dysfunction: results of the 'Cologne Male Survey'. Int J Impot Res. 2000 Dec;12(6):305-11. doi: 10.1038/sj.ijir.3900622. PMID 11416833
- [Background] McKinlay JB. The worldwide prevalence and epidemiology of erectile dysfunction. Int J Impot Res. 2000 Oct;12 Suppl 4:S6-S11. doi: 10.1038/sj.ijir.3900567. PMID 11035380
- [Background] Nicolosi A, Glasser DB, Kim SC, Marumo K, Laumann EO; GSSAB Investigators' Group. Sexual behaviour and dysfunction and help-seeking patterns in adults aged 40-80 years in the urban population of Asian countries. BJU Int. 2005 Mar;95(4):609-14. doi: 10.1111/j.1464-410X.2005.05348.x. PMID 15705089
- [Background] Yee CH, Chan ES, Hou SS, Ng CF. Extracorporeal shockwave therapy in the treatment of erectile dysfunction: a prospective, randomized, double-blinded, placebo controlled study. Int J Urol. 2014 Oct;21(10):1041-5. doi: 10.1111/iju.12506. Epub 2014 Jun 17. PMID 24942563
- [Background] Zhao C, Kim SW, Yang DY, Kim JJ, Park NC, Lee SW, Paick JS, Ahn TY, Moon KH, Chung WS, Min KS, Suh JK, Hyun JS, Park K, Park JK. Efficacy and safety of avanafil for treating erectile dysfunction: results of a multicentre, randomized, double-blind, placebo-controlled trial. BJU Int. 2012 Dec;110(11):1801-6. doi: 10.1111/j.1464-410X.2012.11095.x. Epub 2012 Mar 27. PMID 22448738
- [Background] Vardi Y, Appel B, Kilchevsky A, Gruenwald I. Does low intensity extracorporeal shock wave therapy have a physiological effect on erectile function? Short-term results of a randomized, double-blind, sham controlled study. J Urol. 2012 May;187(5):1769-75. doi: 10.1016/j.juro.2011.12.117. Epub 2012 Mar 15. PMID 22425129
- [Background] Vardi Y, Appel B, Jacob G, Massarwi O, Gruenwald I. Can low-intensity extracorporeal shockwave therapy improve erectile function? A 6-month follow-up pilot study in patients with organic erectile dysfunction. Eur Urol. 2010 Aug;58(2):243-8. doi: 10.1016/j.eururo.2010.04.004. Epub 2010 May 6. PMID 20451317
- [Background] Feldman HA, Goldstein I, Hatzichristou DG, Krane RJ, McKinlay JB. Impotence and its medical and psychosocial correlates: results of the Massachusetts Male Aging Study. J Urol. 1994 Jan;151(1):54-61. doi: 10.1016/s0022-5347(17)34871-1. PMID 8254833
- [Background] Gruenwald I, Appel B, Vardi Y. Low-intensity extracorporeal shock wave therapy--a novel effective treatment for erectile dysfunction in severe ED patients who respond poorly to PDE5 inhibitor therapy. J Sex Med. 2012 Jan;9(1):259-64. doi: 10.1111/j.1743-6109.2011.02498.x. Epub 2011 Oct 18. PMID 22008059
- [Background] Aicher A, Heeschen C, Sasaki K, Urbich C, Zeiher AM, Dimmeler S. Low-energy shock wave for enhancing recruitment of endothelial progenitor cells: a new modality to increase efficacy of cell therapy in chronic hind limb ischemia. Circulation. 2006 Dec 19;114(25):2823-30. doi: 10.1161/CIRCULATIONAHA.106.628623. Epub 2006 Dec 4. PMID 17145991
- [Background] Lei H, Liu J, Li H, Wang L, Xu Y, Tian W, Lin G, Xin Z. Low-intensity shock wave therapy and its application to erectile dysfunction. World J Mens Health. 2013 Dec;31(3):208-14. doi: 10.5534/wjmh.2013.31.3.208. Epub 2013 Dec 24. PMID 24459653